CLINICAL TRIAL: NCT05997199
Title: The Effect of Serum Vitamin D on the Recovery Rate of Bell Palsy
Brief Title: The Effect Vitamin D on the Recovery Rate of Bell Palsy
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Özlem Kaleoğlu, MD, Principle Investigator, Umraniye Education and Research Hospital
Other Study IDs: B.10.1.THK.4.34.H.GP.0.01/76
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Bell Palsy; Vitamin D Deficiency; Facial Paralysis
MeSH Terms: conditions — Bell Palsy; Vitamin D Deficiency; Facial Paralysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients with vitamin D deficiency and having Vitamin D Replacement
  Interventions: Dietary Supplement: Vitamin D replacement
- Group 2: Control Group. Patients with vitamin D deficiency but not getting Vitamin D replacement

INTERVENTIONS:
Dietary Supplement: Vitamin D replacement — Group 1 with vitamin D deficiency will be getting a standart vitamin D replacement of 50.000 IU/week for 8 weeks.
  Groups: Group 1

SUMMARY:
Patients aged between 18-65 who visit the Physical Medicine and Rehabilitation outpatient clinic diagnosed with Bell Palsy will be included in the study. The patients' Bell Palsy grade will be evaluated by Houseman Brahman (HB) Scale and their disability level will be evaluated by Facial Disability Index (FDI). Their serum vitamin D level will be noted. The patients having vitamin D deficiency will be randomized into two groups. Group 1 will be given 50.000 IU/week vitamin D replacement for 8 weeks. All the patients will be included in a standard physical therapy and home exercise program. Both groups will be asked for a control visit at weeks 8.Their clinical recovery will be evaluated by HB staging and FDI by the Physical Medicine and Rehabilitation specialist who is blind to the randomization.

DETAILED DESCRIPTION:
Patients aged between 18-65 who visit the Physical Medicine and Rehabilitation outpatient clinic diagnosed with Bell Palsy will be included in the study. Facial palsy stages of patients will be graded from 1 to 6 according to the Houseman Brahman (HB) staging system. In order to determine the disability criteria of the patients, a form called Facial Disability Index (FDI)-Facial Disability Index will be filled. This scale consists of 10 questions and is a validated test evaluating the physical and social function of the patient. The patients having vitamin D deficiency will be randomized into two groups. One group will be getting a vitamin d replacement treatment for 8 weeks. A physical therapy program in the form of a standard exercise program including electrical stimulation and facial paralysis exercises will be organized for all the patients. The patients will be evaluated at 8th week by HB and FDI.

ELIGIBILITY:
Inclusion Criteria:

* Being cooperative-orientated
* Willing to participate in the Physical Therapy home exercise program

Exclusion Criteria:

* Being Non cooperative, disorientated
* Failure to comply with the Physical Therapy home exercise program
* History of malignancy
* Additional neurological disease
* Having cranial pathologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed with Bell palsy and treated with standard medical treatment in the last 3 weeks
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Houseman Brahman (HB) Level | HB stages of the patients will be recorded at week 8.
  Facial palsy stages of patients will be graded from 1 to 6 according to the Houseman Brahman (HB) staging system. Grade 1 refers to normal facial nerve function whereas 6 refer to complete paralysis.
Facial Disability Index (FDI) | FDI of the patients will be recorded at week 8.
  This scale consists of 10 questions and is a validated test evaluating the physical and social function of the patient. It is scored out of 100. Higher score is the best result.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Kaleoğlu, M.D, Principal Investigator — Umraniye Education and Research Hospital
Locations (1):
- Özlem Kaleoğlu, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No